CLINICAL TRIAL: NCT07141472
Title: Effects of a Glucagon-like Peptide-1 (GLP-1) Booster™ on Blood Glucose, HbA1c, Insulin, Glucagon, GLP-1, GIP, and Amylin Levels, Body Weight and Body Fat in Overweight Adult Men and Women
Brief Title: Glucagon Like Peptide 1 (GLP-1) Booster™ RCT Study
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawry Han (Industry)
Responsible Party: Sponsor-Investigator, Lawry Han, Principal Investigator, Alpine Biotech LLC
Organization: Alpine Biotech LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB20241210H
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Blood Sugar; High; Overweight and Obesity; Fat Loss; GLP-1; Glucagon
Keywords: GLP-1; blood glucose; HbA1c; insulin; glucagon; GIP; Amylin
MeSH Terms: conditions — Hyperglycemia; Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group who take GB (Experimental): GLP-1 Booster (GB) is a composition designed to increase the endogenous production of GLP-1, improve the activity of GLP-1, enhance the body's response to GLP-1, and thus eventually help people reduce glucose, suppress food intake and lose body fat. GB contains Green tea (Camellia sinensis) leaf extract, Gardeniae (Gardenia jasminoides Ellis) fructus extract, Turmeric (Curcuma longa) root extract, Black pepper (Piper nigrum) extract,Fenugreek (Trigonella foenum-graecum) seed extract, Ginseng (Panax ginseng) root extract, and White kidney bean (Phaseolus vulgaris) extract. Each of these ingredients has been commonly consumed by humans as food sources or supplements and thus has an undebatable safety profile.
  Interventions: Dietary Supplement: GB
- Placebo Group (Placebo Comparator): Placebo is a product that resemble Active product but does not contain any of the active ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GB — GLP-1 Booster (GB) is a composition designed to increase the endogenous production of GLP-1, improve the activity of GLP-1, enhance the body's response to GLP-1, and thus eventually help people reduce glucose, suppress food intake and lose body fat. GB contains Green tea (Camellia sinensis) leaf extract, Gardeniae (Gardenia jasminoides Ellis) fructus extract, Turmeric (Curcuma longa) root extract, Black pepper (Piper nigrum) extract,Fenugreek (Trigonella foenum-graecum) seed extract, Ginseng (Panax ginseng) root extract, and White kidney bean (Phaseolus vulgaris) extract. Each of these ingredients has been commonly consumed by humans as food sources or supplements and thus has an undebatable safety profile.
  Arms: Active Group who take GB
Dietary Supplement: Placebo — Placebo is a product that resemble active GB but does not contain any of the active ingredients
  Arms: Placebo Group

SUMMARY:
BACKGROUND GLP1 booster (GB) was designed to stimulate the endogenous production of GLP1, which in turn releases insulin, controls blood glucose level, suppresses appetite and thus helps people lose weight.

PURPOSE In prior study, GB was clinically shown to reduce blood sugar level, increase GLP-1 production, and help body fat loss. The purpose of this RCT study is to further assess several clinical endpoints and questionnaires in healthy volunteers taking the new GB formula vs placebo, in the hope of confirming the efficacy and safety of GB.

SCOPE The scope of this protocol covers the non-clinical portion as well as the assessment of several clinical endpoints and questionnaires. In brief, this study is a randomized controlled clinical trial for a total of 26 weeks. Data analysis will involve measuring the clinical endpoints across the group at different timepoints (week 0, 13 and 26).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be over the age of 18.
* Volunteers cannot be smokers.
* Volunteers cannot be currently taking a dietary supplement or prescription for weight loss.
* Exercising volunteers must maintain their regimen consistently throughout the course of the 26-week study.
* Caffeine drinking volunteers must maintain their caffeine intake consistently throughout the course of the 26-week study.
* Volunteers need to be overweight but not obese, as defined by having a BMI between 25.0 and 29.9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
fasting blood HbA1c level | 26 weeks
  lab
fasting blood glucose level | 26 weeks
  lab
fasting blood insulin level | 26 weeks
  lab
fasting blood GLP-1 level | 26 week
  lab
fasting blood glucagon level | 26 weeks
  lab
fasting blood GIP level | 26 weeks
  lab
fasting blood Amylin level | 26 weeks
  lab
fasting body weight | 26 weeks
  measurement
body fat mass | 26 week
  measurement
waist hip ratio | 26 weeks
  measurement

SECONDARY OUTCOMES:
satiety score | 26 weeks
  questionnaire measuring satiety level from 1 - 10; the higher the score, the more satiety.
resting metabolic rate | 26 weeks
  measurement
Blood pressure | 26 weeks
  both systolic and diastolic pressures
Heart rate | 26 weeks
  measurement
Energy level | 26 weeks
  questionnaire measuring energy level from 1 - 10; the higher the score, the more energy.

CONTACTS AND LOCATIONS:
Overall Officials: Lawry Han, PhD, Principal Investigator — Alpine Biotech
Locations (1):
- Alpine Bio, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No